CLINICAL TRIAL: NCT05667051
Title: Endocan Biomarker Level in Gingival Crevicular Fluid in Periodontitis Patients With Type 2 Diabetes Mellitus [A Comparative Cross-Sectional Study]
Brief Title: Endocan Biomarker Level in Gingival Crevicular Fluid in Periodontitis Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Emad Ayad, MSc candidate, Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology Department, Faculty of Dentistry, Alexandria University, Alexandria University
Other Study IDs: #256
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Periodontitis; Diabetes Mellitus
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlled type 2 diabetes mellitus
- Diabetes mellitus free patients

SUMMARY:
Aim of the current study was to evaluate Endocan biomarker level in gingival crevicular fluid of patients with stage 1 or 2 (mild to moderate) periodontitis with controlled type 2 diabetes mellitus (DM) and compare it to that in DM free periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Probing pocket depths (PPD) ≤ 5 mm.
* Clinical attachment level (CAL) ≤ 4 mm.
* Type 2 DM, for at least the past 3 years.
* HbA1c ≤ 7%.

Exclusion Criteria:

* Uncontrolled Diabetes Mellitus.
* Systemic antibiotic or anti-inflammatory medication use in the previous 2 months.
* Non-surgical periodontal therapy in the previous 6 months.
* Surgical periodontal therapy in the previous 12 months.
* Use of calcium channel blockers, phenytoin, or cyclosporine.
* Pregnancy.
* Smokers

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 1 or 2 (mild to moderate) periodontitis having ≤ 4 mm attachment loss at least in one site were included in the study these were divided into two groups, with controlled type 2 diabetes mellitus, and systemically healthy stage 1 or 2 (mild to moderate) periodontitis patients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Endocan level | Day 1
  Endocan level in gingival crevicular samples was assessed by commercially available ELISA kit (Bioneovan Co., Ltd, Elisa Human Endocan/esm-1 ELISA Kit. Beijing, China). Assays were performed according to the manufacturer's instructions. Color change will be measured with a microplate reader (Hellma GmbH & Co. KG. Müllheim, Germany) at 450 nm. Concentrations were determined based on the respective assay standard curve. All samples were run in duplicate and values will be averaged
Pocket probing depth (PPD) | Day 1
  PPD was assessed at six different sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) per tooth at all teeth present, except third molars. PPD was assessed using Williams calibrated periodontal probe and recordings were made to the nearest mm; observations close to 0.5 mm were rounded to the upper whole mm.
Clinical Attachment Level (CAL) | Day 1
  CAL was assessed at six different sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) per tooth at all teeth present, except third molars. CAL was assessed using Williams calibrated periodontal probe and recordings were made to the nearest mm; observations close to 0.5 mm were rounded to the upper whole mm.
Percentage of bleeding on probing sites (BOP%) | Day 1
  BOP% was assessed at six different sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) per tooth at all teeth present, except third molars. BOP% was assessed using Williams calibrated periodontal probe and the number of sites with BOP were divided by the total number of examined sites and multiplied by 100 to calculate the percentage

CONTACTS AND LOCATIONS:
Overall Officials: Emad Ayyad, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Maha Abou Khadr, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Mona Ayyad, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt; Gillan El-Kimary, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt